CLINICAL TRIAL: NCT04296552
Title: Study Protocol of the Bergen Brain-gut-microbiota-axis Study: a Prospective Case-report Characterization and Dietary Intervention Study to Evaluate the Effects of Microbiota Alterations on Cognition and Anatomical and Functional Brain Connectivity in Patients With Irritable Bowel Syndrome
Brief Title: Brain-Gut-Microbiota Interaction in IBS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Haukeland University Hospital (Other)
Collaborators: National Research Council, Spain (Other Government); Genetic Analysis AS (Unknown); Lovisenberg Diakonale Hospital (Other); University of Bergen (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2015-01621
Record Dates: First submitted 2020-03-04; First posted 2020-03-05 (Actual); Last update posted 2020-06-30 (Actual); Status verified 2020-06

CONDITIONS: Irritable Bowel Syndrome; Functional Gastrointestinal Disorders
MeSH Terms: conditions — Irritable Bowel Syndrome; Gastrointestinal Diseases

STUDY DESIGN:
Intervention Model Description: The study is an open, single-centre, case-control characterisation study, followed by open label dietary intervention for a subgroup of subjects with IBS-D. Exploratory trial.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- 12 week lowFODMAP dietary intervention (Experimental): Patients with IBS-D are enrolled in a 12 week strict lowFODMAP dietary intervention study.
  Interventions: Other: Dietary lowFODMAP intervention

INTERVENTIONS:
Other: Dietary lowFODMAP intervention — Twelve week strict lowFODMAP dietary intervention, involving restricted intake of fermentable carbohydrates (FODMAPs).

SUMMARY:
Are you what you eat? How can dietary components influence microbial composition of the gut and function of the peripheral and central nervous system? The gut and brain is linked through complex mechanisms of sensorimotor functions of the immune system, the hypothalamic-pituitary-adrenal-axis, the enteric nervous system and microbiota.

In this project, a multitude of factors contributing to the bidirectional neurobiological communication along the brain-but-axis will be investigated. No disease of the brain-gut axis has been elucidated, therefore our investigations involves approaching a large span of components and processes involved in the axis. This study is carried out as a case-report study (baseline, IBS n=100, healthy controls n=40) followed by a dietary intervention (IBS-D n=60). Through multivariate analyses, the investigators will identify patterns of factors contributing to patient symptomatology and pathology, followed by big data analysis leading to stratification of sub-classification of irritable bowel syndrome (IBS).

DETAILED DESCRIPTION:
Data from deep phenotype characterization of 100 patients with IBS and 40 healthy age (between 18 and 65) and gender-matched controls will be collected between May 2019 and December 2021. Psychometric tests, questionnaires, biological samples (blood, faeces, saliva and GI biopsies from antrum, duodenum and sigmoid colon), assessment of gastric accommodation and emptying using transabdominal ultrasound, vagal activity, and functional and structural magnetic resonance imaging (MRI) of the brain, will be carried out. A subgroup of 60 patients with IBS-D will be further included in a 12-week low Fermentable Oligo-, Di-, Mono-saccharides And Polyols (FODMAP) dietary intervention-study to determine short and long-term effects of diet on symptoms, microbiota composition, molecular GI signatures, cognition and behavioural traits, and structural and functional brain signatures. Deep machine learning, prediction tools and big data analysis will be used for multivariate analysis allowing disease stratification and diagnostic biomarker detection.

ELIGIBILITY:
Inclusion Criteria:

* Subject must be between 18 and 65 years of age
* Fulfil the ROME-IV criteria for IBS

  1. Had recurrent abdominal pain on average at least 1 day per week during the previous 3 months that is associated with alterations in bowel habits.
  2. Duration at least six months.

Exclusion Criteria:

* Pharmacological treatment affecting the GI-tract, including treatment for depression
* Organic disease:

  1. coeliac disease
  2. inflammatory bowel disease
  3. neurological diseases
  4. diabetes
  5. active helicobacter pylori infection
  6. polycystic ovary syndrome
* Treated with systemic antibiotics within the last 3 months
* Use painkillers regularly, other than paracetamol
* Pregnant
* Previous intestinal surgery (appendectomy is OK)
* Claustrophobic or have metallic implants that are not MR compatible
* Vegan or vegetarian
* Been travelling outside Europe within the last three weeks (or plan to travel in the nearest future)
* Probiotics or lowFODMAP-diet within the last three weeks
* Participation in any other simultaneous clinical study
* Inability to comprehend and respond to questionnaires or follow dietary guidance

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2019-05-20 (Actual); Primary Completion 2021-12-31 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Short-term dietary lowFODMAP responder will be measured using IBS-symptom severity score | At 4 weeks
  A minimum of 50 point reduction in IBS-symptom severity score (range 0-500: mild (75-175), moderate (175-300) and severe (>300), below 75 (remission))
Long-term dietary lowFODMAP responder will be measured using the IBS-symptom severity score | At 12 weeks
  A minimum 50 point reduction in IBS-symptom severity score (range 0-500: mild (75-175), moderate (175-300) and severe (>300), below 75 (remission))

CONTACTS AND LOCATIONS:
Locations (1):
- Haukeland University Hospital, Bergen, Vestlandet, Norway

IPD SHARING:
Plan to Share IPD: Yes
De-identified stool samples, blood chemistry and symptom severity scores will be shared with collaborators.
Supporting Information: Study Protocol
Time Frame: The data will become available post microbiota-analysis until the end of the study period.

REFERENCES:
- [Derived] Bjorkevoll SMG, Randulff Hillestad EM, Lied GA, Teige ES, Steinsvik EK, Berentsen B, Lundervold AJ. A 12-Week Strict Low FODMAP Diet Reduces the Severity Levels of Fatigue, Depression, Anxiety, and Inattention in Patients with Irritable Bowel Syndrome. Curr Dev Nutr. 2025 Jun 6;9(7):107483. doi: 10.1016/j.cdnut.2025.107483. eCollection 2025 Jul. PMID 40654377
- [Derived] Lundervold AJ, Billing JE, Berentsen B, Lied GA, Steinsvik EK, Hausken T, Lundervold A. Decoding IBS: a machine learning approach to psychological distress and gut-brain interaction. BMC Gastroenterol. 2024 Aug 15;24(1):267. doi: 10.1186/s12876-024-03355-z. PMID 39148020
- [Derived] Berentsen B, Nagaraja BH, Teige EP, Lied GA, Lundervold AJ, Lundervold K, Steinsvik EK, Hillestad ER, Valeur J, Bronstad I, Gilja OH, Osnes B, Hatlebakk JG, Haasz J, Labus J, Gupta A, Mayer EA, Benitez-Paez A, Sanz Y, Lundervold A, Hausken T. Study protocol of the Bergen brain-gut-microbiota-axis study: A prospective case-report characterization and dietary intervention study to evaluate the effects of microbiota alterations on cognition and anatomical and functional brain connectivity in patients with irritable bowel syndrome. Medicine (Baltimore). 2020 Sep 11;99(37):e21950. doi: 10.1097/MD.0000000000021950. PMID 32925728